CLINICAL TRIAL: NCT00722176
Title: A Six-Week, Randomized, Double-Blind, Parallel Group Extension Study To Evaluate The Long-Term Safety, Tolerability, And Efficacy Of Low And High Doses Of Bl-1020 Compared To Risperidone
Brief Title: Extension Study To Evaluate The Long-Term Safety, Tolerability, And Efficacy Of Low And High Doses Of Bl-1020
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: BioLineRx, BioLineRx
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BL-1020 IIb (Extension)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — perphenazine GABA ester; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): BL-1020 10 mg
  Interventions: Drug: BL-1020
- 2 (Experimental): BL-1020 10-30 mg
  Interventions: Drug: BL-1020 10-30 mg
- 3 (Active Comparator): risperidone
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: BL-1020 — 10 mg
  Arms: 1
Drug: BL-1020 10-30 mg — BL-1020 10-30 mg
  Other Names: BL-1020 High Dose
  Arms: 2
Drug: risperidone — risperidone
  Arms: 3

SUMMARY:
A Six-Week, Randomized, Double-Blind, Parallel Group Extension Study To Evaluate The Long-Term Safety, Tolerability, And Efficacy Of Low And High Doses Of Bl-1020 Compared To Risperidone, In Schizophrenic Patients Previously Treated In Study Bl-1020 Iib For A Maximum Of Six Weeks With Bl-1020 (High Dose, Low Dose), Risperidone Or Placebo

DETAILED DESCRIPTION:
This is a six-week, randomized, double blind, multi-center, parallel group Extension to the BL-1020 IIb study. In this Extension Study in patients hospitalized with schizophrenia who were previously treated in the BL-1020 IIb study with BL-1020 (low dose: 10 mg/day; high dose: target dose 30 mg/day), risperidone (target dose: 8 mg/day) or placebo after experiencing an acute exacerbation of schizophrenia. Patients who completed the 6 week treatment period and/or all efficacy assessments in Study BL-1020 IIb are eligible to continue double-blind treatment in this optional 6 week Extension Study. Approximately 220 patients will be enrolled in this study: Treatment Group IE (n=82, 10 mg/day BL-1020); Treatment Group IIE (n=82: target dose 30 mg/day BL-1020); Treatment Group IIIE (n=55; target dose 8 mg/day risperidone). Study drug (BL-1020 or risperidone) will be administered orally, once daily, in a doubleblinded manner, during this six-week Extension Study

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years of age at the time of entry into the BL-1020 IIb study
2. Has provided informed consent to participate in the Extension Study
3. Has completed 6 weeks of treatment and/or completed all efficacy assessments in Study BL-1020 IIb
4. Females must have negative serum pregnancy test, or be post-menopausal, or if fecund, must practice established methods of birth control (oral contraceptive tablets, hormonal implant device, hormone patch, injectable contraceptive, intrauterine device [IUD]) for at least two months prior to screening
5. Females must use an established method of birth control (as above) AND a barrier method (condom, diaphragm, contraceptive foam) while taking study medication
6. Has a caregiver or an identified responsible person (e.g., family member, social worker, nurse) who will support him/her to ensure compliance with the treatment and outpatient visits
7. Is willing to comply with not taking any prohibited medications during participation in the study
8. Successful completion of End of Study assessments from BL-1020 IIb

Exclusion Criteria:

1. Is unwilling or unable to provide informed consent
2. Is unwilling or unable, in the opinion of the Investigator, to comply with study instructions
3. Has a medical condition that would put him/her at risk for continuing in the study
4. Score > 9 on Modified InterSePT Scale for Suicidal Thinking (Modified ISST)
5. Tested positive for drugs of abuse during the initial 6 weeks of treatment (Study BL-1020 IIb)
6. Has been non-compliant with the study medication dosing and/or study procedures during the initial 6 weeks of treatment in Study BL-1020 IIb
7. Is judged by the PI to be inappropriate for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
changes from baseline in vital signs, laboratory and ECG evaluations, physical/neurological examination, Extrapyramidal Symptom Rating Scale (ESRS), and incidence of adverse events (AEs) and adverse drop-outs (ADOs). | 6 weeks

SECONDARY OUTCOMES:
Comparisons between each of the BL-1020 treatment groups and the risperidone group | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Knisevich, MD, Principal Investigator — University Hills Clinical Research
Locations (1):
- University of California, Irvine, Irvine, California, United States